CLINICAL TRIAL: NCT05169294
Title: The Effect of Fine Motor Skills Training Through Telerehabilitation on Handwriting, Occupational Performance, Fine Motor Skills and Hand Skills in Children With Diplegic Cerebral Palsy
Brief Title: The Effect of Fine Motor Skills Training Through Telerehabilitation in Children With Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ekin Akpınar (Other)
Responsible Party: Sponsor-Investigator, Ekin Akpınar, Occupational Therapist, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KA20090
Record Dates: First submitted 2021-12-13; First posted 2021-12-23 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Diplegia, Spastic
Keywords: cerebral palsy; handwriting; occupational therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Children to be included in the study will be divided into intervention (n: 30) and control (n: 30) groups by randomization. Block randomization will be done using randomizer.org. Children in both groups will be given an occupational therapy home program for intervention goals.
  Children in the intervention group will be given telerehabilitation and fine motor skills training for a total of 8 weeks, 45 minutes a day, 3 days a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Telerehabilitation Program; Other: Written Home Program
- Control (Active Comparator)
  Interventions: Other: Written Home Program

INTERVENTIONS:
Other: Telerehabilitation Program — Telerehabilitation program: Intervention will be applied by video interview for eight weeks, 3 days a week, 45 minutes a day through the Zoom application. The application is free and can be installed on desktop or laptop computers, tablets and smartphones. The content of the activities to be done for that session by phone call to the parent before the interventions; Information will be given about the preparations such as keeping the materials on the table, suitable environment for that week's session and camera angle. Instructions and tips for parent support during the intervention will be given before and during the session. Intervention will be focused on fine motor skills, handwriting skills and activities of daily life of the individuals.
  Arms: Intervention
Other: Written Home Program — Home program: After the evaluations, the activities towards the determined goals will be communicated to the parents as a home program in written and electronic format. Instructions and key points for the correct implementation of the activities will be presented to the parent, both in writing and verbally; The parent will be able to send questions and receive feedback to the therapists over the phone at any stage of the eight-week home program intervention process. No intervention will be applied to the child through direct video calls.

SUMMARY:
The aim of this study is to compare the effect of occupational therapy intervention through two-way video call, versus occupational therapy home program in written form; on handwriting skills, occupational performance, fine motor and hand skills in children with diplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with diplegic cerebral palsy
* Being between the ages of 7-12
* Being able to read and write
* To be at level I-III in the Manual Ability Classification System (MACS)
* To have the necessary devices (phone, tablet or computer) for video calling
* Not being able to come to the faculty to conduct the first evaluation face to face
* Not receiving occupational therapy in any special education center

Exclusion Criteria:

* Presence of another neurological and/or psychiatric disease
* Not giving consent to the study Individuals included in the study will be randomly assigned to the intervention and control groups. It is planned to keep the number of individuals in the intervention and control groups equal.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Children's Hand Skills (ACHS) | 8 weeks
  ACHS is an observational assessment that measures the effectiveness of manual dexterity in children aged 2-12 years when participating in meaningful activities. Scoring items are categorized as: manual gestures, body-related dexterity, arm-hand use, adaptive dexterity hand use, general quality, and bimanual skills. A six-level Likert scale is used to score all skill items (Chien, Brown, & McDonald, 2010; Chien et al, 2011; Chien & Brown, 2012). The application of this test takes about 10 minutes.
Minnesota Handwriting Assessment | 8 weeks
  The Minnesota Handwriting Assessment is a writing quality assessment that includes copying seven words containing all the letters of the alphabet (Guzman Pasculli, Hiraga, & Pellegrini, 2017). Evaluation scores six components of the text: speed, legibility, form, alignment, size and spacing (Alhussaini. Meram & Buragada, 2016). The Turkish adaptation, validity and reliability of the Minnesota Handwriting Assessment was performed by Kavak and Bumin (Kavak & Bumin, 2006). This assessment takes less than 5 minutes to apply.
Shriners Hospital Upper Extremity Evaluation (SHUEE) | 8 weeks
  SHUEE is an assessment developed to measure upper extremity function in children with hemiplegic cerebral palsy. SHUEE is a video-based assessment administered by an occupational therapist using standardized objects and tasks. The evaluation takes about 15 minutes and is then scored by the occupational therapist (Davids, Piece, Wagner et al, 2006). Turkish validity and reliability of SHUEE was done by Bumin et al. (Bumin, Özsezen, & Yıldız, 2018).
Bruininks-Oseretsky Test of Motor Proficency 2- Short Form (BOT-2 SF) | 8 weeks
  BOT-2 is a tool that is frequently used in the evaluation of psychomotor characteristics in individuals aged 4-21 years (Jirovec, Musalek, & Mess, 2019).
  It is available in two versions, full form and short form. Four areas of psychomotor characteristics can be measured with BOT-2: (1) fine manual control, (2) accuracy and integrity, (3) manual coordination, and (4) physical coordination (Jirovec et al, 2019).
  In our study:
  * Item 2 of the bilateral coordination subtest,
  * Item 3, 4, 5 and 8 of the visual motor control subtest
  * Item 7 of the upper extremity speed and motion accuracy subtest, will be applied and scored.
  The application of these substances takes approximately 5 minutes. Since BOT-2 is a motor assessment test, there is no need for a Turkish validity and reliability study to be performed.
Canadian Occupational Performance Measure | 8 weeks
  COPM is a client-centered assessment tool used in occupational therapy (Carswell, McColl, Baptiste et al, 2004; Harris & Eng, 2004; Parker & Sykes, 2006; Enemark Larsen, Jessen Winge, & Christensen, 2019) The COPM assessment helps individuals to identify, prioritize and evaluate their occupational performance difficulties (Law, Baptiste, Carswell et al, 2015; Enemark Larsen et al, 2019). The Turkish adaptation, validity and reliability of the COPM were made by Torpil et al. (Torpil, Ekici, & Bumin, 2017). This assessment will take approximately 20 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided